CLINICAL TRIAL: NCT07005011
Title: Comparison of the Efficacy of the Oral Irrigator Versus Interdental Brushes in the Oral Hygiene of Patients With Gingivitis: a Randomised Study
Brief Title: Comparison of the Efficacy of Oral Irrigator Versus Interdental Brushes in the Oral Hygiene of Patients With Gingivitis: a Randomised Study
Acronym: Hydro-Paro
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024_RIPH_30_Hydro-Paro
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Gingivitis
Keywords: Gingivitis; oral irrigator; interdental brushes; interdental hygiene
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: "oral irrigator" group (Experimental): group 1: patients using oral irrigator as interdental hygiene tools
  Interventions: Other: oral irrigator
- group2: "calibrated interdental brushes" group (Active Comparator): group 2: patients using calibrated interdental brushes as interdental hygiene tools
  Interventions: Other: oral irrigator

INTERVENTIONS:
Other: oral irrigator — oral irrigator

SUMMARY:
Periodontal health is a public health issue because of the frequency of periodontal disease (more than 50% of the French population suffers from severe periodontitis (Bourgeois, Bouchard and Mattout 2007)), its negative impact on patients' quality of life, speech, self-confidence and well-being, and its association with the development of chronic pathologies (diabetes, metabolic syndrome, rheumatoid arthritis, cardiovascular disease).

Gingivitis is a reversible inflammatory disease of the superficial tissues supporting the teeth. If left untreated, this inflammation will become chronic and spread apically to the deep tissues supporting the tooth, evolving into periodontitis with irreversible damage. The aetiopathogenic phenomena that lead to the onset of periodontal disease are complex, but one of the main aetiopathogenic factors is the bacterial biofilm found in the form of dental plaque.

Maintaining correct oral hygiene remains the main means of preventing periodontal disease (Chapple et al. 2018). Plaque control is achieved by the dental surgeon through scaling and resurfacing at intervals appropriate to the patient, but also by the patient themselves. Mechanical removal of plaque by brushing prevents it from accumulating and prevents the onset of these diseases. This control by the patient is essential to the effectiveness of periodontal treatments and the maintenance of periodontal health.

Plaque control by the patient using a toothbrush is not sufficient and must be supplemented by the use of interdental hygiene (Lindhe and Koch 1967). To date, the most effective interdental hygiene tools for reducing gingival inflammation and the plaque index are interdental brushes (Sälzer et al. 2015). However, their effectiveness requires professional calibration to enable adaptation to all sites, which can then reduce patient compliance through the need to use multiple tools.

Oral irrigator were developed in the 1960s and in 2001 the American Academy of Periodontology recognised their value in reducing gingival inflammation. The oral irrigator Sonicare HX8432 Ultra, Philips® was developed recently, combining water and air. Its pulsatile action is considered to be more conservative of gingival soft tissue and qualitatively modifies the composition of dental plaque.

The advantage of this tool is that, unlike interdental brushes, it does not require calibration and is simpler to use.

DETAILED DESCRIPTION:
The main objective of this study was to evaluate the benefit of using oral irrigator Sonicare HX8432 Ultra, Philips® in patients with gingivitis on the reduction of the interproximal plaque index (API, Lange, 1975) after 12 weeks of use compared to the use of calibrated interdental brushes.

The secondary objectives of this study were to assess the benefit of using oral irrigator Sonicare HX8432 Ultra, Philips® in patients with gingivitis compared with using calibrated interdental brushes :

* reduction in the plaque control record (PCR) (O'Lheary et al., 1972) after 12 weeks' use
* reduction in Bleeding on probing (BOP) index (Ainamo & Bay, 1975) after 12 weeks' use
* on improvement in oral health-related quality of life (GOHAI - Geriatric Oral Health Assessment Index) after 12 weeks' use

ELIGIBILITY:
Inclusion Criteria:

* with gingivitis (according to the International Classification of Periodontal Diseases; Chapple et al., 2018 i.e. a BOP greater than 10%).
* with at least 10 pairs of antagonistic teeth
* able to carry out oral hygiene procedures independently
* able to understand the instructions for using interdental devices
* fluent in French
* adults
* affiliated to a social security scheme
* agreeing to take part in the study

Exclusion Criteria:

* daily use of one of the study devices (hydropulper, whatever the model, or calibrated interdental brushes)
* with a medical history that could compromise the protocol (psychiatric, medical or pharmacological disorders such as the use in the week prior to inclusion of anti-inflammatory drugs, antibiotics or any compound that could alter or modify the inflammatory response)
* with eating disorders
* with ongoing orthodontic treatment
* protected by law (guardianship, curatorship, safeguard of justice)
* pregnant or breast-feeding women
* refusing to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Approximal plaque index (API - Lange, 1977) | 12 weeks
  API is the number of interdental spaces covered by plaque divided by the total number of interdental spaces studied, expressed as a percentage. To calculate it, the interdental spaces are visually examined by the dental surgeon to determine whether or not the surface is covered by plaque.

SECONDARY OUTCOMES:
Plaque control record (PCR - O'Lheary et al., 1972) | 12 weeks
  the PCR is the number of plaque-covered tooth surfaces divided by the total number of tooth surfaces studied, expressed as a percentage. To calculate it, the 4 tooth surfaces (vestibular, mesial, distal, lingual) of all the teeth present will be examined by the dental surgeon using a manual periodontal probe and plaque developer to determine whether or not the surface is covered by dental plaque.
Bleeding on probing (BOP - Ainamo et Bay, 1975) | 12 weeks
  BOP is the number of bleeding tooth surfaces divided by the total number of tooth surfaces examined, expressed as a percentage. To calculate it, the 4 tooth faces (vestibular, mesial, distal, lingual) of all teeth present will be examined by the dental surgeon using a manual periodontal probe to determine the presence or absence of bleeding.
General Oral Health Assessment Index (GOHAI - Tubert-Jeanin et al., 2003) | 12 weeks
  The GOHAI consists of 12 questions coded from "never" (5) to "always" (1), covering the last 3 months. The GOHAI score is calculated by adding up the scores for all the questions to obtain a score ranging from 12 to 60. A score of 57 to 60 reflects good oral health quality of life; a score of 51 to 56 reflects average oral health quality of life; and a score below 50 reflects poor oral health quality of life.

IPD SHARING:
Plan to Share IPD: Undecided